CLINICAL TRIAL: NCT05676021
Title: The Effect of Health Education Supported by Motivational Interviewing on the Adherence to Medication of Patients With COVID-19 Diagnosed at Home
Brief Title: The Effect of Motivational Interviewing on the Adherence to Medication of Patients With COVID-19 Diagnosed at Home
Acronym: MOTIVATION
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Saglik Bilimleri Universitesi Gulhane Tip Fakultesi (Other)
Responsible Party: Principal Investigator, Serpil Özdemir, PhD, RN, Saglik Bilimleri Universitesi Gulhane Tip Fakultesi
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: MOTIVATION
Record Dates: First submitted 2022-12-20; First posted 2023-01-09 (Actual); Last update posted 2023-01-09 (Actual); Status verified 2023-01

CONDITIONS: Drug Compliance
Keywords: COVID-19; Medication Compliance; Motivational Interviewing; Health Education
MeSH Terms: conditions — Medication Adherence; COVID-19; Health Education | interventions — Motivational Interviewing

STUDY DESIGN:
Intervention Model Description: randomised control trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention group (Experimental): On the second day of the COVID-19 antiviral drug treatment, the participant assigned to the intervention group was interviewed face-to-face during the home visit by providing isolation measures. In the face-to-face meeting, the "COVID-19 Medication Use Brochure" was given and it was stated that the participants would be video-talked about the topics included in the booklet at an appropriate time on the same day, and time was planned. In the interview, it was decided to allow the participant to tell about their antiviral drug use, to learn about their feelings, thoughts and behaviors about drug use, to reveal their feelings of indecision and anxiety about treatment, to determine their resistance to drug use, to reveal their intrinsic motivation, to support them and to change their behavior. It was intended to take action to advance the cycle of change.
  Interventions: Behavioral: motivational interview
- control group (No Intervention): After randomization, the participants in the control group continued to receive health care according to the standard COVID-19 drug treatment procedures determined by the Ministry of Health. No other intervention was performed apart from the participant standard COVID-19 drug therapy procedures in the control group.

INTERVENTIONS:
Behavioral: motivational interview — motivational interview-based health education
  Arms: intervention group

SUMMARY:
Summary Objective: The aim of this study is to determine the effect of health education supported by motivational interviewing on drug therapy compliance of patients with COVID-19 who are followed at home.

Materials and Methods: 100 participants with a diagnosis of COVID-19 followed at home were divided into intervention (50) and control (50) groups by block randomization method. The data at the beginning of the study were obtained with the Introductory Information Form (16 questions). At the end of the study, the Medication Compliance Notification Scale and the level of satisfaction with medication (1 question) questionnaire were applied to the participants. The "Medicine Calendar" was used to track the drug use status of all participants. In the study, while the control group received standard COVID-19 drug therapy, in addition to the standard treatment to the intervention group; On the second day of the treatment, health education supplemented with motivational interviewing was conducted online.

Results: At the end of the study, it was found that the mean score of drug compliance (16.12±5.37) of the participants in the intervention group was higher than the mean score of the participants in the control group (9.96±5.62) (p<0.05). The mean score of drug compliance (16.12±5.37) of the participants in the intervention group at the end of the study was higher than the mean score at the beginning of the study (11.02±4.03) (p<0.05). The mean adherence score of the control group at the end of the study (9.96±5.62) was found to be lower than the mean score of adherence (11.40±4.93) at the beginning of the study (p<0.05). At the end of the study, when the participants in the intervention group were examined, it was seen that they were higher than the participants in the control group.

Conclusion: At the end of the study; The mean score of the intervention group's medication adherence scale increased significantly compared to the control group receiving standard medication; it was evaluated that this increase did not reach the desired level. This situation revealed how important the motivational interview-based health education given by nurses is in increasing drug compliance.

DETAILED DESCRIPTION:
This study was designed as a randomized controlled trial. Between June 2021 and January 2022, it was carried out at the Gallipoli District Health Directorate, which is affiliated to the Çanakkale Provincial Health Directorate. The eligibility of patients for participation in the study was evaluated by the investigator. The sample size is in line with the results of the study of Çakmak and Kapucu in which they examined the effect of motivational interviewing on drug compliance in patients receiving oral chemotherapy; Assuming Type 1 error α=0.05, Type 2 error β=0.05, effect width f=0.6 ratios, 45 participants in each group in the G*Power program at 90% power and 95% confidence interval. counted as 90 participants. Taking into account possible losses, it was decided to add 10% reserve participants, and a total of 100 participants, 50 in each group, formed the sample size. Standard COVID-19 drug treatment procedures determined by the Ministry of Health are applied to COVID-19 positive patients by the District Health Directorate's filiation team and in the standard COVID-19 drug treatment procedure; On the day of the diagnosis of the disease, phone calls are made with the patients and the medical anamnesis of the patients is taken. On the same day, home visits are made to patients who do not have contraindication to antiviral drugs. In this visit, antiviral drugs are delivered to the patients by the filiation team, explaining how to use the drugs, and the "Favipiravir Usage Brochure" prepared by the Ministry of Health is given to the patients. Patients who were on the first day of treatment, who were determined to be COVID-19 positive, were asked if they volunteered to participate in the study, after a phone call by the principal investigator, followed by a brief briefing about the study, after the call of the filiation team. The condition of meeting the inclusion criteria of the study, excluding the level of drug compliance, of the patients who volunteered to participate in the study was examined. A face-to-face meeting was planned with participants who met the inclusion criteria on the same day. The patients who volunteered to participate in the study were given COVID-19 isolation precautions (overall, N95 and surgical mask, visor and gloves, social distance) and made a home visit at the scheduled time, "Voluntary Consent Forms" were given, and they were received in a sealed envelope to ensure contact isolation. During the face-to-face meeting, all patients were given the "Favipiravir Use Brochure" prepared by the Ministry of Health, explaining how to use the drug, and the "COVID-19 Drug Schedule" follow-up form, and how this form should be filled. Approximately antiviral drugs were delivered to the patient. However, the home visit was terminated by informing the patients that a video phone call would be made on the second day of the treatment.A video phone call was made with all participants on the second day of treatment. First of all, the participants were informed that they would be asked some questions about their personal information and medication, that there was no right or wrong answer option in the questions, and the participants were asked to share the most appropriate answer without hesitation. The questions and answer options in the introductory information form and the Drug Compliance Notification Scale were conveyed to the participant without guidance, and the answers of the participants were recorded. By ending the interview, data on the descriptive characteristics of the participants were collected, and the scores of the drug compliance reporting scale were evaluated. After the initial evaluation, patients with a mean drug adherence score above 20 (n=124) were excluded from the study. At this stage, randomization was achieved by assigning the participants to the intervention and control groups using the double-block randomization method according to the order of the case date.

ELIGIBILITY:
Inclusion Criteria:

* Those who volunteered to participate in the study
* 18 years old and over,
* Able to read and write Turkish,
* Having a COVID-19 patient followed at home,
* Having the equipment to make video calls over the internet connection,
* Individuals with a drug compliance reporting scale score below 20 points

Exclusion Criteria:

* Contraindicated to use antiviral drug (Favipiravir) (liver failure, kidney failure, active chemotherapy treatment)
* Pregnant,
* Patients who were hospitalized for any reason during the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2021-06-15 (Actual); Primary Completion 2021-12-20 (Actual); Study Completion 2022-01-20 (Actual)

PRIMARY OUTCOMES:
drug compliance reporting scale mean score | 5 days
  The Drug Compliance Reporting Scale is a Likert-type scale consisting of 5 items. The score to be taken from the scale is between 5 and 25. An increase in the scale score is interpreted as an increase in the level of drug compliance.

SECONDARY OUTCOMES:
increased drug compliance | 5 days
  The cut-off score of the drug compliance reporting scale is 20 points. At the end of the study, participants who score 20 points or more from the scale are considered to have a high level of drug compliance.

CONTACTS AND LOCATIONS:
Overall Officials: burcu yılmaz, Principal Investigator — Ministry of Health
Locations (1):
- University of Health Sciences, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No